CLINICAL TRIAL: NCT04761783
Title: BESPOKE Study of ctDNA Guided Immunotherapy
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-043-NCP
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Melanoma; Non-small Cell Lung Cancer
Keywords: BESPOKE; circulating tumor DNA
MeSH Terms: conditions — Colorectal Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — There are two arms to this study: A prospective arm that will enroll 1539 patients, and a historical control (retrospective arm) that will enroll 513 patients.
  Each participant in the Prospective arm will have received the commercially available SIGNATERA™ test.
  Subjects prospectively enrolled and whom consent to "Optional future Research" may have bio-specimens stored for future research. The historical arm (retrospective cohort) will not have any bio-specimens collected or stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective arm: Patients will receive SIGNATERA™ test results and the immunotherapy treatment regimen, dosing schedule, duration of treatment, number of cycles, and modifications during treatment will be at the discretion of the HCP. Patients will be followed for up to two years with periodic whole blood collection. Treatment administered, disease-free survival, overall survival, time to recurrence, physician questionnaires and patient-reported outcomes will be recorded.
- Control arm: Control cases must have undergone immunotherapy treatment and have follow-up data available in their medical record at the participating site for two years following initiation of immunotherapy or death.

SUMMARY:
This is a prospective data collection study of patients with advanced solid tumors who will receive standard of care immunotherapy (IO) and will be monitored with SIGNATERA™ testing. SIGNATERA™ test will be performed at baseline and during routine care. The test results will be part of assessing tumor response. The correlation between SIGNATERA™ test results and subsequent treatment decisions will be examined to compare actual treatment delivered against treatment decisions potentially impacted by SIGNATERA™ results. Treatment administered, tumor assessment results, time to progression, overall survival, physician questionnaires, and patient-reported outcomes will be collected/recorded.

DETAILED DESCRIPTION:
Primary Objective:

● To examine the impact of SIGNATERA™ on clinical decision-making regarding continuation, discontinuation, escalation, or de-escalation of immunotherapy.

Secondary Objective:

● To prospectively evaluate the utility of SIGNATERA™ as a tool to detect early evidence of response or progression in patients with advanced solid tumors receiving immune checkpoint inhibitors.

ELIGIBILITY:
Prospective Inclusion Criteria:

1. Male or female patients 18 years of age or older at the time of signing informed consent form (ICF)
2. Any patient with documented metastatic or locally advanced, unresectable cancer of the types within the following cohorts:

   1. Melanoma
   2. Non-small cell lung cancer
   3. Colorectal cancer
3. Patients must be clinically eligible and planned to receive therapy with an anti-neoplastic agent that works by immune checkpoint blockade, anti-PD-1, anti-CTLA-4, or anti-PD-L1:

   1. Pembrolizumab (Keytruda)
   2. Nivolumab (Opdivo)
   3. Ipilimumab (Yervoy)
   4. Durvalumab (Imfinzi)
   5. Cemiplimab (Libtayo)
   6. Atezolizumab (Tecentriq)
   7. Avelumab (Bavencio)
4. Patients must have measurable disease according to RECIST criteria, and at least one lesion that can be accurately measured in at least one dimension as >10 mm.
5. Patients must be able to follow study visit schedule and willing to provide up to 20 mL of peripheral blood samples at the indicated time points
6. ECOG Performance status 0,1, or 2
7. Able to read, understand and provide written informed consent
8. Willing and able to comply with the study requirements
9. Selected by their HCP to receive SIGNATERA testing according to the current evidence-informed schedule as part of their routine of practice

Prospective Exclusion Criteria:

1. Female patients that are pregnant
2. History of bone marrow or organ transplant
3. Medical condition that would place the patient at risk as a result of blood donation, such as bleeding disorder
4. Serious medical condition that may adversely affect ability to participate in the study
5. Has initiated Immunotherapy

Control Arm Inclusion Criteria:

1. Male or female patients 18 years of age or older at the time of signing informed consent form (ICF)
2. Any patient with documented metastatic or locally advanced, unresectable cancer of the types within the following cohorts:

   1. Melanoma
   2. Non-small cell lung cancer
   3. Colorectal cancer
3. Patients must be clinically eligible and planned to receive therapy with an anti-neoplastic agent that works by immune checkpoint blockade, anti-PD-1, anti-CTLA-4, or anti-PD-L1:

   1. Pembrolizumab (Keytruda)
   2. Nivolumab (Opdivo)
   3. Ipilimumab (Yervoy)
   4. Durvalumab (Imfinzi)
   5. Cemiplimab (Libtayo)
   6. Atezolizumab (Tecentriq)
   7. Avelumab (Bavencio)
4. Patients must have measurable disease according to RECIST criteria, and at least one lesion that can be accurately measured in at least one dimension as >10 mm.
5. Patients must be able to follow study visit schedule and willing to provide up to 20 mL of peripheral blood samples at the indicated time points
6. ECOG Performance status 0,1, or 2
7. Able to read, understand and provide written informed consent
8. Willing and able to comply with the study requirements
9. Selected by their HCP to receive SIGNATERA testing according to the current evidence-informed schedule as part of their routine of practice

Control Arm Exclusion Criteria:

1. Female patients that are pregnant
2. History of bone marrow or organ transplant
3. Medical condition that would place the patient at risk as a result of blood donation, such as bleeding disorder
4. Serious medical condition that may adversely affect ability to participate in the study
5. Has initiated Immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with advanced colorectal cancer, non-small cell lung cancer, or melanoma
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Examine the impact of SIGNATERA on treatment decisions on tumor assessment timepoints after initiation of immunotherapy | 2 years
  Percent of patients who have their immunotherapy treatment regimen changed due to post-treatment SIGNATERA ctDNA test result

SECONDARY OUTCOMES:
To determine progression free survival according to ctDNA change | 2 years
  Compare progression free survival, defined as the duration of time between enrollment and an increase in severity of disease as determined by patient's treating physician, between groups determined by change in ctDNA
Determine overall survival according to ctDNA change | 2 years
  Compare overall survival, defined as the duration of time between enrollment and death for any reason, between groups determined by change in ctDNA
Determine response rate according to ctDNA change in cases with progression of disease on first or second tumor assessment and who continue treatment. | 2 years
  Compare percentage of patients that experience partial or complete response during the study, between groups determined by change in ctDNA
To determine progression free survival according to ctDNA change in cases who achieve stable disease on first tumor assessment. | 2 years
  Compare progression free survival between groups determined by change in ctDNA
To determine duration of response according to ctDNA change in cases who achieve partial response or complete response as best overall response. | 2 years
  Compare duration of response, defined as the length of time from initial response to disease progression, between groups determined by change in ctDNA
To determine percentage of patients with at least 6 months of durable clinical response according to ctDNA change in patients who achieve at least partial response on best tumor assessment. | 2 years
  Among all patients that are clinically identified to experience partial or complete response, percentage that have at least 6 months durable clinical response as determined by ctDNA change
Determine the impact of SIGNATERA on the confidence in immunotherapy treatment decisions based on the number of patients in which treating physician reports SIGNATERA made them more confident in immunotherapy treatment regimen | 2 years
  Percent of patients whose treating physician reported that SIGNATERA result made them more confident in selected immunotherapy treatment regimen
Determine the impact of SIGNATERA in informing immunotherapy treatment decisions | 2 years
  Percent of patients whose immunotherapy treatment regimen was changed as a result of SIGNATERA and/or whose treating physician reported that SIGNATERA result made them more confident in selected immunotherapy treatment regimen
Determine the impact of SIGNATERA on patient reported outcomes | 2 years
  Assess patient anxiety levels and wellbeing in patients receiving SIGNATERA ctDNA test results.
  Patient responses to patient reported outcome questionnaires:
  EORTC QLQ-C30
  Assess if SIGNATERA makes patients feel that they are receiving the right treatment and determine if patients will continue to use Signatera in the future to monitor their cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Aleshin, MD, Principal Investigator — Natera, Inc.
Locations (1):
- Natera, San Carlos, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kasi PM, Chakrabarti S, Sawyer S, Krainock M, Poklepovic A, Ansstas G, Maninder M, Malhotra M, Ensor J, Gao L, Eroglu Z, Ellers S, Billings P, Rodriguez A, Aleshin A. BESPOKE IO protocol: a multicentre, prospective observational study evaluating the utility of ctDNA in guiding immunotherapy in patients with advanced solid tumours. BMJ Open. 2022 May 30;12(5):e060342. doi: 10.1136/bmjopen-2021-060342. PMID 35636789